CLINICAL TRIAL: NCT04797936
Title: A Randomized, Open-label, Multicentre, Comparative Study of Therapeutic Efficacy, Safety, and Tolerability of BNO 1030 Extract, in the Treatment of Mild Forms of COVID-19
Brief Title: BNO 1030 Extract (Imupret) in the Treatment of Mild Forms of COVID-19
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ivano-Frankivsk National Medical University (Other)
Responsible Party: Principal Investigator, Vasyl Popovych, Head of department "Otolaringology, children otolaryngology and surdology", Ivano-Frankivsk National Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BERI_UA_IMU_2020_000003751
Record Dates: First submitted 2021-03-08; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Covid19; Nasopharyngitis; Anosmia; Fever; Myalgia; Cough; Nasal Congestion
MeSH Terms: conditions — COVID-19; Nasopharyngitis; Anosmia; Fever; Myalgia; Cough; Nasal Obstruction | interventions — imupret; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group BNO 1030 (Active Comparator): BNO 1030
  Interventions: Drug: BNO 1030
- Control group (Other): Standard care
  Interventions: Other: Standard care

INTERVENTIONS:
Drug: BNO 1030 — Imupret 25 drops х 6 times per day for 14 days
  Other Names: Imupret
  Arms: Treatment group BNO 1030
Other: Standard care — isolation mode symptomatic therapy as needed: antipyretic (paracetamol) saline solutions in the nose x 4 times a day -14 days
  Arms: Control group

SUMMARY:
According to WHO (World Health Organisation) data, about 40% of patients with COVID-19 (Corona Virus SARS-CoV-2) have a mild course of the disease, namely, cases of mild course are of great danger from the point of view of the spread of infection, since the main source of infection is a sick person. The mild course of COVID-19 is characterized by a number of nonspecific symptoms: fever, cough, sore throat, nasal congestion, malaise, headache, muscle pain. Evidence has emerged of loss of smell as a symptom of COVID-19 infection. Anosmia/hyposmia in the absence of other respiratory diseases, such as allergic rhinitis, acute rhinosinusitis, or chronic rhinosinusitis, are considered as a clinical marker of COVID-19 infection in a pandemic.For people with a mild course of the disease, WHO recommends providing home care, and the recommendations come down to observing a sanitary-hygienic regimen and taking antipyretics if necessary. Unfortunately, the treatment of patients with a mild course is still outside the interest of medical science. In its updated strategy to curb the spread of COVID-19, WHO states the need for diagnosis, effective isolation, and treatment of patients with mild to moderate severity of the clinical course of patients.Currently, there is experience with the use of the drug Imupret for the treatment of nasopharyngitis associated with other viral pathogens, in particular Epstein-Barr virus. It was shown that the use of a Phyto preparation helps to accelerate the regression of symptoms characteristic of nasopharyngitis, as well as accelerate the elimination of the virus from the body. Obviously, the proven activity of Imupret is important in relation to the activation of factors of nonspecific immunity, which is important in confronting viruses, including COVID-19. Another obvious factor that is important for the treatment of viral diseases is the synergism of the active substances in oak bark and walnut leaves with respect to inhibition of reverse transcriptase of a wide range of respiratory viruses, as well as the anti-inflammatory effect of the drug. Confirmation of the therapeutic effect of Imupret for the treatment of nasopharyngitis associated with COVID-19 would allow the development of new therapeutic tools to combat this infection and put into practice updated WHO emphasis on national health systems: it is important to identify, treat and isolate all cases of COVID-19, including cases with mild or moderate severity of the disease.

DETAILED DESCRIPTION:
The new coronavirus (2019-nCoV) from Wuhan is currently of great concern, as the virus is spreading rapidly around the world and the number of cases and deaths is constantly growing. The main cause of death is the severe course of COVID-19 disease, which includes pneumonia, acute respiratory distress syndrome (ARDS), sepsis, and septic shock. As the spread of COVID-19 is progressing worldwide, the focus is on the rapid identification, testing, and treatment of patients with severe COVID-19 and the hospitalization of people with the highest risk of fatal outcomes.

Less attention is paid to cases of mild disease. According to WHO data, about 40% of patients with COVID-19 have a mild course of the disease, namely, cases of mild course are of great danger from the point of view of the spread of infection, since the main source of infection is a sick person. An infected person, even with minor clinical symptoms, can infect between 1.5 and 3.5 people and spread the virus among approximately 368 people in just five infection cycles. The mild course of COVID-19 is characterized by a number of nonspecific symptoms: fever, cough, sore throat, nasal congestion, malaise, headache, muscle pain. Evidence has emerged of loss of smell as a symptom of COVID-19 infection. South Korea, China, and Italy have already proven that a significant number of patients with proven COVID-19 infection developed anosmia/hyposmia. In Germany, more than 2 out of 3 confirmed cases are reported to have anosmia. Anosmia/hyposmia in the absence of other respiratory diseases, such as allergic rhinitis, acute rhinosinusitis, or chronic rhinosinusitis, are considered as a clinical marker of COVID-19 infection in a pandemic.

For people with a mild course of the disease, WHO recommends providing home care, and the recommendations come down to observing a sanitary-hygienic regimen and taking antipyretics if necessary. Unfortunately, the treatment of patients with a mild course is still outside the interest of medical science. However, in its updated strategy to curb the spread of COVID-19, WHO states the need for diagnosis, effective isolation, and treatment of patients with mild to moderate severity of the clinical course of patients.

Fever, cough, sore throat, nasal congestion, malaise, headache, muscle pain, and decreased sense of smell are typical symptoms of acute nasopharyngitis. It is believed that the previously described coronaviruses account for 10-15% of cases of nasopharyngitis, so it is not surprising that the new COVID-19 virus can also cause anosmia in infected patients. These patients need isolation and treatment because they are covert carriers that contribute to the rapid spread of COVID-19.

Currently, there is experience with the use of the drug Imupret for the treatment of nasopharyngitis associated with other viral pathogens, in particular Epstein-Barr virus. It was shown that the use of a Phyto preparation helps to accelerate the regression of symptoms characteristic of nasopharyngitis, as well as accelerate the elimination of the virus from the body. Obviously, the proven activity of Imupret is important in relation to the activation of factors of nonspecific immunity, which is important in confronting viruses, including COVID-19. Another obvious factor that is important for the treatment of viral diseases is the synergism of the active substances in oak bark and walnut leaves with respect to inhibition of reverse transcriptase of a wide range of respiratory viruses, as well as the anti-inflammatory effect of the drug. Confirmation of the therapeutic effect of Imupret for the treatment of nasopharyngitis associated with COVID-19 would allow the development of new therapeutic tools to combat this infection and put into practice updated WHO emphasis on national health systems: it is important to identify, treat and isolate all cases of COVID-19, including cases with mild or moderate severity of the disease.

ELIGIBILITY:
Inclusion Criteria:

Age 18-70 years old;

* Clinical signs of a mild form of COVID-19 (acute nasopharyngitis associated with 2019-nCoV), assessed by direct contact or remotely: sudden onset, fever, cough

  + at least one of the following:
  * nasal congestion;
  * discharge from the nose (front and back rhinorrhea);
  * anosmia/hyposmia;
* Contact with a confirmed or suspected case of COVID-19
* The possibility of treatment on an outpatient basis subject to the self-isolation mode

Exclusion Criteria:

Indications for inpatient treatment

* The presence of immunodeficiency conditions, oncological diseases, chronic diseases of the cardiovascular or broncho-pulmonary system, diabetes mellitus.
* Individual intolerance to the components of the drug.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-12-19 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
Day of response to treatment from baseline to end of treatment (up to two weeks) - decrease in the average score of the symptom assessed by the patient (VAS, 0-10 points for each symptom) by 50% compared to baseline. | Visit 1 (Day 1), Visit 2 (Day 4), Visit 3 (Day 14)
  patient's assessment of the symptoms 11 Point visual analogue scale 0 - absent symptom, 10 - the maximum severity of the symptom) for rhinorrhea, nasal congestion, rhinolalia, anosmia, sore throat, general condition, fever.

SECONDARY OUTCOMES:
Symptom Dynamics (assessed by patients) | Every day in the treatment phase up to 14 days
  Symptom measurement by patient's self assessment (General condition, sore throat, fever, rhinorrhea, cough, nasal congestion via ten-point visual analogue scale (VAS, 0 - 10 points (0- no symptom; 10 -maximal expression of the symptom).

OTHER OUTCOMES:
Symptom Dynamics (assessed by docktor) | At Visit 1 (Day 0) and at Visit 3 (day 14)
  Symptom measurement by doctors (General condition, sore throat, fever, rhinorrhea, cough, nasal congestion via 5-point criteria: 0-4 points/symptom. 0 - none symptom; 1- mild; 2- moderate; 3- severe; 4- very severe).

CONTACTS AND LOCATIONS:
Overall Officials: Vasyl Popovych, Professor, Principal Investigator — Ivano-Frankivsk National Medical University
Locations (1):
- Ivano-Frankivsk National Medical University, Ivano-Frankivsk, Ukraine

IPD SHARING:
Plan to Share IPD: No